CLINICAL TRIAL: NCT05271604
Title: A Phase 2 Open-Label Study of Ozuriftamab Vedotin (BA3021) in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Phase 2 Open Label Study of BA3021 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA3021-002
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of Head and Neck; Recurrent Squamous Cell Carcinoma of the Head and Neck; Metastatic Cancer; Metastatic Squamous Cell Carcinoma of the Head and Neck
Keywords: Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort M1 (Experimental): Monotherapy BA3021 Q2W dosing regimen
  Interventions: Biological: Ozuriftamab Vedotin
- Cohort M2 (Experimental): Monotherapy BA3021 2Q3W dosing regimen
  Interventions: Biological: Ozuriftamab Vedotin
- Cohort N1 (Experimental): Neoadjuvant/induction setting combination therapy of BA3021 2Q3W dosing regimen, pembrolizumab Q3W dosing regimen, and BA3071 Q3W dosing regimen prior to surgery.
  Interventions: Biological: Ozuriftamab Vedotin; Biological: Pembrolizumab; Biological: Evalstotug (BA3071)
- Cohort C1 (Experimental): Combination therapy of BA3021 2Q3W dosing regimen, pembrolizumab Q3W dosing regimen, and BA3071 Q3W dosing regimen
  Interventions: Biological: Ozuriftamab Vedotin; Biological: Pembrolizumab; Biological: Evalstotug (BA3071)
- Cohort C2 (Experimental): Combination therapy of BA3021 2Q3W dosing regimen, and pembrolizumab Q3W dosing regimen
  Interventions: Biological: Ozuriftamab Vedotin; Biological: Pembrolizumab
- Cohort C3 (Experimental): Combination therapy of BA3021 2Q3W dosing regimen and cetuximab QW dosing regimen
  Interventions: Biological: Ozuriftamab Vedotin; Biological: Cetuximab

INTERVENTIONS:
Biological: Ozuriftamab Vedotin — Conditionally active biologic anti-ROR2 antibody drug conjugate
Biological: Pembrolizumab — PD-1 inhibitor
  Arms: Cohort C1; Cohort C2; Cohort N1
Biological: Evalstotug (BA3071) — Conditionally active biologic anti-CTLA-4 checkpoint blockade antibody
  Arms: Cohort C1; Cohort N1
Biological: Cetuximab — Epidermal growth factor receptor (EGFR) antagonist
  Other Names: Erbitux
  Arms: Cohort C3

SUMMARY:
This is a multi-center, open-label Phase 2 study designed to evaluate the efficacy and safety of BA3021 as monotherapy and combination therapy in patients with recurrent or metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx. Patients may not have a primary tumor site of nasopharynx (any histology).
* Neoadjuvant/induction setting (Cohort N1): Patient with newly diagnosed Stage III SCCHN who are eligible for induction therapy with resectable tumors. No prior treatments, including surgery, radiation, or systemic treatment, for SCCHN are allowed.
* Recurrent or metastatic setting: Histologically or cytologically confirmed recurrent or metastatic SCCHN Stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
* First-line - Combination Cohorts (C1 and C2): Patients must have NO prior systemic therapy administered in the locally recurrent or metastatic setting. Previous treatments with PD-1/L1 inhibitor or anti-CTLA-4 treatment are not allowed.
* Second-line (Combination Cohort C3) and Second-line+ (Monotherapy Cohorts M1 and M2): Patients must have documented treatment failure of no more than one approved PD-1/L1 inhibitor either administered alone or in combination.

Patients must have measurable disease.

* Age ≥ 18 years
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as well as known or suspected allergy or intolerance to any agent given during this study.
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) per RECIST v1.1 | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR according to RECIST v1.1
Incidence of Adverse Events or Serious Adverse Events as assessed by CTCAE v5 | Up to 24 months
  Measured by frequency and severity of adverse events as assessed by CTCAE v5

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 24 months
  Time from the first documented OR until the first documented disease progression or death (due to any cause), whichever occurs first
Progression-free survival (PFS) | Up to 24 months
  Time from the first dose of IP until the first documentation of disease progression or death due to any cause, whichever occurs first.
Best overall response (BOR) | Up to 24 months
  All post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy
Disease control rate (DCR) | Up to 24 months
  Proportion of patients with a best overall response of confirmed CR, confirmed PR, or stable disease (SD) ≥ 12 weeks.
Time to response (TTR) | Up to 24 months
  Time from the first dose of investigational product until the first documentation of OR.
Overall survival (OS) | Up to 24 months
  Time from the first dose of BA3021 treatment until death due to any cause.
Complete response (CR) | Up to 24 months
  Proportion of patients with a best overall response of confirmed CR

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Christiana Care Helen Graham Cancer Center, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Washington University Medical Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah